CLINICAL TRIAL: NCT05090657
Title: Bacterial Eradication of the Nasal Epithelium From Infectious Toxins With PDT (BENEFIT-PDT)
Brief Title: Nasal Photodisinfection in All Patients Presenting for Surgery for a Wide Range of Surgical Procedures
Acronym: BENEFIT-PDT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ondine Biomedical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BENEFIT-PDT 01
Record Dates: First submitted 2021-10-10; First posted 2021-10-25 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Surgical Site Infections; Nosocomial Infection; Healthcare Associated Infections
Keywords: Staphylococcus aureus; Photodynamic therapy; Photodisinfection; Methylene blue; Nasal decolonization; Surgical infections
MeSH Terms: conditions — Surgical Wound Infection; Cross Infection; Staphylococcal Infections | interventions — Methylene Blue; chlorhexidine gluconate; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Intervention Model Description: The sample size will be one month of all surgical cases and is estimated at 500-600 cases. Both genders and a wide range of ages and medical conditions will be represented from all ethnic/demographic groups and of varying health status.
Masking Description: As an infection prevention study the intervention of nasal photodisinfection will be applied to all willing participants within the time frame. Pre and post intervention nasal cultures will be performed. Clinicians will not be aware of these results during the patients hospital course.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Open label presurgical nasal decolonization (Other): All patients presenting for surgery will be offered nasal decolonization with the combination product. After informed consent a nasal culture will be obtained followed by a 4-minute nasal decolonization treatment and a post-treatment culture. The intervention consists of swabbing the nose with a methylene blue/chlorhexidine gluconate solution followed by non-thermal nasal illumination with red light. There will only be a single treatment.
  Interventions: Combination Product: methylene blue 0.01%/chlorhexidine gluconate 0.25% + light activation

INTERVENTIONS:
Combination Product: methylene blue 0.01%/chlorhexidine gluconate 0.25% + light activation — After topical application photosensitive solution bilateral nasal light diffusers will be inserted into each nostril and two 2-minute non-thermal light applications of 670 nm light will be used to activate the photosensitizer to achieve an oxidative burst to destroy pathogens.
  Other Names: photodisinfection (PD), photodynamic therapy (PDT), photoactivated chemotherapy (PACT),

SUMMARY:
This is a Phase 2 single-center, open-label, single-arm, study of a microbiological endpoint using antimicrobial photodynamic therapy (aPDT) for nasal disinfection in all patients (universal) presenting for surgery at an acute care hospital for a wide range of surgical procedures.

DETAILED DESCRIPTION:
The purpose of the proposed study is to gather data regarding the safety and efficacy of nasal photodisinfection treatment in eliminating colonization of the anterior nares with S. aureus. The anterior nares are often considered the primary reservoir of S. aureus and other pathogens on the body, therefore, this product could play an important role in helping to eliminate this pathogen reservoir in patients. Since photodisinfection is a non-antibiotic approach that does not generate antibiotic resistance, this could be a beneficial approach to achieving nasal disinfection. Additionally, photodisinfection has an extremely broad spectrum of activity and is effective against bacterial, viral, and fungal pathogens including emerging pathogens such as C. auris.

This is a Phase 2 study. Nasal cultures will be performed on all patients admitted for surgery at Memorial Health University Medical Center over a 1-month period. This will determine the prevalence rate of S. aureus and other pathogens in community patients who are being admitted for surgery. The results of this culture will not be known to the research staff until several days later. Clinical trial subjects will universally receive a nasal disinfection treatment followed by a post-treatment culture. This will demonstrate the efficacy of nasal disinfection against Staphylococcus aureus and methicillin-resistant Staphylococcus aureus.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form within 30 days of surgery.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female ≥ 18 years of age.
4. Patient being admitted for a surgical procedure.
5. Ability to tolerate a 4-minute non-painful nasal light illumination.

Exclusion Criteria:

1. Male or female <18 years of age.
2. Inability to tolerate insertion of the nasal light illuminator due to nares size, shape, or anatomical variants.
3. Known allergic reactions to components of the nasal disinfection treatment including methylene blue or chlorhexidine gluconate.
4. Nasal obstructions precluding placement of light illuminator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-08-06 (Actual); Study Completion 2022-08-06 (Actual)

PRIMARY OUTCOMES:
Microbiological efficacy | Within 1 hour of start of surgery
  All pre-surgical subjects will be screened by plate culture for Staphylococcus aureus nasal carriage. All subjects will receive the nasal decolonization treatment and then be screened again for Staphylococcus aureus carriage.
Side effects of nasal photodisinfection | 30 days
  Subjects will be evaluated for any treatment related side effects including rhinorrhea, mucosal irritation, laryngeal irritation, sneezing or any reported adverse event.

SECONDARY OUTCOMES:
Incidence of surgical site infections | 30 days
  Patients will be followed up for any reported post-operative infections

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A. Thacker, MD, Principal Investigator — Memorial University Medical Center, Savannah, GA
Locations (1):
- Memorial University Medical Center, Savannah, Georgia, United States

IPD SHARING:
Plan to Share IPD: No